CLINICAL TRIAL: NCT07357740
Title: A Phase 2 Study to Compare Two Presentations of CagriSema in Participants With Type 2 Diabetes
Brief Title: A Research Study to Compare Two Different Versions of Injectable CagriSema in People With Type 2 Diabetes
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9388-8468; U1111-1323-3766 (Other: World Health Organization (WHO)); 2025-522570-37 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2026-01-21; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CagriSema in device 1 + Placebo CagriSema B in device 2 (Experimental): Participants will receive CagriSema in device 1 followed by placebo matched to CagriSema B in device 2 subcutaneously once weekly in a dose escalation manner.
  Interventions: Drug: CagriSema; Drug: Placebo CagriSema
- CagriSema B in device 2 + Placebo CagriSema in device 1 (Experimental): Participants will receive CagriSema B in device 2 followed by placebo matched to CagriSema in device 1 subcutaneously once weekly in a dose escalation manner.
  Interventions: Drug: CagriSema; Drug: Placebo CagriSema

INTERVENTIONS:
Drug: CagriSema — Cagrilintide and Semaglutide will be administered subcutaneously using device 1 or device 2.
Drug: Placebo CagriSema — Placebo matched to Cagrilintide and Placebo matched to Semaglutide will be administered subcutaneously using device 1 or device 2.

SUMMARY:
This study is being done to look at how well a study medicine called CagriSema helps people with diabetes lower their blood sugar. In this study the sponsor will compare two version of CagriSema injected by two different types of injection devices. Which treatment participants get is decided by chance. CagriSema is still being tested in studies and is not yet available for doctors to prescribe. The study will last for about 38 weeks.

ELIGIBILITY:
Inclusion Criteria

* Male or female (sex assigned at birth, inclusive of all gender identities).
* Age 18-64 years (both inclusive) at the time of signing the informed consent.
* Diagnosed with type 2 diabetes mellitus greater than or equal to (>=) 180 days before screening.
* Glycated haemoglobin (HbA1c) 7.0-10.5 percent (%) (53-91 [millimoles per mole] mmol/mol) (both inclusive) as determined by the central laboratory at screening.
* Stable daily dose >= 90 days before screening of metformin at effective or maximum tolerated dose as judged by the investigator.
* Body mass index (BMI) between 25.0 and 39.9 kilograms per square metre (kg/m^2) (both inclusive) at screening. BMI will be calculated in the electronic case report form (eCRF) based on height and body weight at screening.

Exclusion Criteria:

* Renal impairment with estimated Glomerular Filtration Rate (eGFR) < 30 millilitre per minute per 1.73 square metre (mL/min/1.73 m^2) as determined by the central laboratory at screening.
* Treatment with any anti-diabetic or anti-obesity medication (irrespective of indication) other than stated in the inclusion criteria within 90 days before screening.
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by an eye examination performed within 90 days before screening or in the period between screening and randomisation.
* Previous exposure to CagriSema in a clinical study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-08-27 (Estimated); Primary Completion 2027-08-25 (Estimated); Study Completion 2027-10-13 (Estimated)

PRIMARY OUTCOMES:
Change in glycated haemoglobin (HbA1c) | Baseline to week 28
  Measured as percentage-points (%-points).

SECONDARY OUTCOMES:
Weekly average cagrilintide (total) and semaglutide concentration (Cavg) based on population pharmacokinetic analyses | From baseline to week 28
  Measured in nanomoles per litre (nmol/L).
Change in HbA1c | From baseline to week 28
  Measured as %-points.
Number of Treatment Emergent Adverse Events (TEAEs) | From baseline to week 35
  Measured as count of events.
Number of clinically significant hypoglycaemic episodes (level 2) (less than [<] 3.0 millimoles per litre [mmol/L]), confirmed by blood glucose (BG) meter, or severe hypoglycaemic episodes (level 3) | From baseline to week 35
  Measured as count of episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (9):
- Denmark (4):
  - Sanos Clinic - Gandrup, Gandrup
  - Sanos Clinic - Herlev, Herlev
  - Sanos Clinic - Vejle, Vejle
  - Regionshospitalet Viborg - Karkirurgisk Afsnit, Viborg
- Slovakia (5):
  - Diakom, spol. s r.o., Poprad
  - MED-DIA CENTRUM s.r.o., Považská Bystrica
  - DIALIPID, s.r.o., Prešov
  - iDia s. r. o., Žiar nad Hronom
  - MEDIVASA, s.r.o., Diabetologicka ambulancia, Žilina

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com